CLINICAL TRIAL: NCT02337673
Title: Screening of Postoperative Pulmonary Complications by Electrical Impedance Tomography in Intensive Care Patients Undergoing Epigastric Surgery
Brief Title: Screening of Postoperative Pulmonary Complications by Electrical Impedance Tomography
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Dr. med. Michael Schuster, Dr. med., Johannes Gutenberg University Mainz
Other Study IDs: JohannesGU-EIT-01
Record Dates: First submitted 2014-05-24; First posted 2015-01-14 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Pulmonary Disease; Postoperative Respiratory Complications; Malignant Neoplasm of Stomach; Liver Diseases; Pancreatic Diseases
Keywords: Postoperative Pulmonary Complication; Electrical Impedance Tomography; Splenectomy; Gastric surgery; Gastrectomy; Pancreatic surgery; Pancreatectomy; Liver surgery; Hemihepatectomy; Cholecystectomy; Acute Respiratory Distress Syndrome; Hypoxemia; Atelectasis; Pulmonary obstruction; Pneumonia; Pneumothorax; Pleural effusion; Pulmonary edema
MeSH Terms: conditions — Lung Diseases; Stomach Neoplasms; Liver Diseases; Pancreatic Diseases; Respiratory Distress Syndrome; Hypoxia; Pulmonary Atelectasis; Airway Obstruction; Pneumonia; Pneumothorax; Pleural Effusion; Pulmonary Edema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether Electrical Impedance Tomography can be used as sensitive and specific predictor in the detection of postoperative pulmonary complications (e.g. pneumonia, bronchitis, acute respiratory distress syndrome, pleural effusion, pneumothorax, pulmonary edema, atelectasis, pulmonary embolism, hypoxemia, hypercapnia, spasms and obstructions of the airway) in patients undergoing epigastric surgery.

DETAILED DESCRIPTION:
* Study cycle:

  1. Check of criteria of inclusion/exclusion
  2. Informed consent
  3. Recording preoperative data via paper case report form
  4. Preoperative EIT measurement
  5. Postoperative EIT measurement
  6. Recording postoperative data via paper case report form

     Patients therapy and any diagnostic investigation during hospital stay (apart from EIT measurement) are performed appropriate to patients individual clinical needs and are independent from participation in this clinical trial. As PPC may result from surgical complications (e.g. intra- /postoperative bleeding, anastomotic leak, infection of the wound, injury of neighboring organs) they are monitored.
* Statistical analysis:

Sample size:

After consultation of Johannes-Gutenberg-University Institute of Medical Biometry and Epidemiology the following procedure was developed: Pre-analysis with 20 patients, then determination of definitive sample size (advised 80 patients).

Population:

Any registered patient is included in population even if no study-treatment was performed. To fulfill Pre-Protocol-Population-criteria EIT-measurement has to be performed before and after elective epigastric surgery and information about PPC must be revealable from patients medical file/records.

* Analysis of efficacy:

  1. Primary objective:

     (A) Incidence of any PPC (postoperative pulmonary complication) until postoperative day 7; Acquisition of PPC might require diagnostic investigation during hospital stay; investigations are only performed appropriate to patients individual clinical needs. As PPC are defined:
     * I: desaturation, increased oxygen demand (data from electronic health record)
     * II: dys-/atelectasis, pleural effusion, pneumothorax, pulmonary vein congestion (data from thoracic x-ray)
     * III: detected respiratory infection/pneumonia, pulmonary edema, Aspiration, non-invasive/CPAP-Ventilation, necessity of pleural drain/of bronchoscopy (data from electronic health record, x-ray)
     * IV: Reintubation (data from electronic health record), ARDS (according to Berlin Definition)

     (B) regional Distribution of Ventilation (Analysis of EIT raw data pre- and postoperative in 4 regions of interest: ventral, mid-ventral, mid-dorsal, dorsal; correlation between PPC and difference in regional Distribution of Ventilation at defined moment)
  2. Secondary objective: post-hoc Analysis (see down Secondary Outcome Measure)

     Average, Median, Quartile, Standard Deviation are detected and shown in Box-plots (type of graphic). Explorative comparison of parameters is effected by t-Test, Mann-Whitney-U-Test, Fisher-Test dependent on normal distribution.
* Quality assurance and data management Design, execution and analyzation of the study is ICH-GCP-conform (Good-Clinical-Practice-Guideline of the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use). All responsible persons are obliged to good clinical practice. All changes in study protocol are to be authorized by responsible Ethics Committee. The P.I. is responsible for source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources (e.g., medical records, paper or electronic case report forms).

Prior to written informed consent all patients are to be informed about character and consequences of the study. With their signature patients permit collection and use of source data. Every patient receives an Identification code for pseudonymization of data. Analyzation and publication of data is effected anonymously only. Data collection is mainly provided in an electronic data base, besides in a paper-based Case Report Form. All electronic and paper-based data and archived in our Clinical Research Center and are accessible for authorized persons (Monitor, Auditor). The study protocol does not provide audits.

Amendment after Pre-analysis:

We conducted a preliminary study of 23 patients for sample size calculation, aligned with the goal of predicting probability of relevant PPC. Power calculation was based on the assumption that 50 % of patients would develop relevant PPC. We performed a power analysis using the Wilcoxon test. The assumption was that AUC of EIT-parameters for distinguishing PPC-affected patients from non-affected patients would be at least 0.65. In order to demonstrate that AUC is indeed above 0.5, a Wilcoxon test can be applied. AUC=0.65 translates into P(X<Y)=0.65. To demonstrate this at the 5%-significance level with a power of 80%, 116 patients are needed. Considering that approximately 10% of patients may not be evaluable, a total sample size of 130 patients was determined. Interim analysis revealed, that incidence of relevant PPC in the study cohort was lower than assumed in sample size calculation. Therefore a higher sample size was necessary than expected. Furthermore, recruiting was slow. We therefore switched from a confirmatory to a descriptive approach.

ELIGIBILITY:
Inclusion Criteria:

* age > 17 years
* no participation in another trial
* mental and physical state allow written consent
* elective epigastric surgery by laparotomy in general anesthesia (e.g. gastrectomy, splenectomy, pancreatic surgery, liver surgery/hemihepatectomy, cholecystectomy)

Exclusion Criteria:

* age < 18 years
* in women: pregnancy
* missing or disability for giving written consent
* emergency patients
* patients after cardiac surgery less than 3 months ago
* patients after pulmonary lobectomy during lifetime
* patients with cardiac stimulator/defibrillator or any other implant with electric activity
* patients with cutaneous lesions or bandage in the area of EIT electrode placement
* patients with instability of the spine
* body mass index > 50

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of a primary care clinic (university hospital) undergoing elective epigastric surgery by laparotomy in general anesthesia with elective postoperative intensive care surveillance.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change of regional ventilation partition (ROI analysis in 8 pulmonary ROIs) from preoperative to postoperative state. | 1.) First EIT-measure: Preoperative Day; 2.) Second EIT-measure: Day of Operation (after extubation) or in between Postoperative Day 1-7 (in case of deferred extubation)
  Comparison of the changed regional ventilation partition to the occurence of postoperative pulmonary complications => calculation of sensitivity and specifity of the primary outcome measure to predict PPC. Statistical analysis: receiver operating characteristic (ROC curve).

SECONDARY OUTCOMES:
Postoperative EIT-measured regional ventilation distribution (ROI analysis in 8 pulmonary ROIs) | 1 week
  Sensitivity and specifiy for appearance of PPC (Postoperative Pulmonary Complications) within Postoperative Day 1-7.
  Statistical analysis: Sensitivity, Specificity, ROC-curve
Postoperative EIT-measured regional ventilation distribution (ROI analysis in 8 pulmonary ROIs) | 1 week
  Correlation of pre-existing pathologic pulmonary conditions with specific postoperative changes in regional distribution of lung ventilation and perfusion assessed by EIT Statistical analysis: Sensitivity, Specificity, ROC-curve
Appearance of all specific forms of PPC (Postoperative Pulmonary Complications) within postoperative day 1-7 | 1 week
  Appearance of all different forms of PPC within Postoperative Day 1-7 and relation to postoperative EIT-measure (ROI analysis in 8 pulmonary ROIs).
  Statistical analysis: Sensitivity, Specificity, ROC-curve
Outcome (e.g. mortality, time of intensive care therapy, ventilator-obligatory-free days on Postoperative Day 1-7 Postoperative EIT-measure is predictive for patients outcome | 1 week
  Sensitivity and specifity of postoperative EIT-measure for mortality. Statistical analysis: Sensitivity, Specificity, ROC-curve
Time of intensive care therapy | 1 week
  Sensitivity and specifity of postoperative EIT-measure for time of intensive care therapy.
  Statistical analysis: Sensitivity, Specificity, ROC-curve
Ventilator-obligatory-free days | 1 week
  Sensitivity and specifity of postoperative EIT-measure for Ventilator-obligatory-free days.
  Statistical analysis: Sensitivity, Specificity, ROC-curve

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bodenstein, Principal Investigator — marc-bodenstein@gmx.de
Locations (1):
- Universitätsmedizin Mainz, Klinik für Anästhesiologie (University Hospital of Johannes Gutenberg-University Mainz, Department of Anesthesiology), Mainz, Rheinland-Pfalz (Rhineland-Palatinate), Germany

REFERENCES:
- [Background] Bodenstein M, David M, Markstaller K. Principles of electrical impedance tomography and its clinical application. Crit Care Med. 2009 Feb;37(2):713-24. doi: 10.1097/CCM.0b013e3181958d2f. PMID 19114889
- [Background] Bodenstein M, Boehme S, Bierschock S, Vogt A, David M, Markstaller K. Determination of respiratory gas flow by electrical impedance tomography in an animal model of mechanical ventilation. BMC Pulm Med. 2014 Apr 29;14:73. doi: 10.1186/1471-2466-14-73. PMID 24779960
- [Background] Hinz J, Neumann P, Dudykevych T, Andersson LG, Wrigge H, Burchardi H, Hedenstierna G. Regional ventilation by electrical impedance tomography: a comparison with ventilation scintigraphy in pigs. Chest. 2003 Jul;124(1):314-22. doi: 10.1378/chest.124.1.314. PMID 12853539
- [Background] Richard JC, Pouzot C, Gros A, Tourevieille C, Lebars D, Lavenne F, Frerichs I, Guerin C. Electrical impedance tomography compared to positron emission tomography for the measurement of regional lung ventilation: an experimental study. Crit Care. 2009;13(3):R82. doi: 10.1186/cc7900. Epub 2009 May 29. PMID 19480694
- [Background] Victorino JA, Borges JB, Okamoto VN, Matos GF, Tucci MR, Caramez MP, Tanaka H, Sipmann FS, Santos DC, Barbas CS, Carvalho CR, Amato MB. Imbalances in regional lung ventilation: a validation study on electrical impedance tomography. Am J Respir Crit Care Med. 2004 Apr 1;169(7):791-800. doi: 10.1164/rccm.200301-133OC. Epub 2003 Dec 23. PMID 14693669